CLINICAL TRIAL: NCT04003636
Title: A Phase 3 Randomized, Double Blind Study of Pembrolizumab Plus Gemcitabine/Cisplatin Versus Placebo Plus Gemcitabine/Cisplatin as First-Line Therapy in Participants With Advanced and/or Unresectable Biliary Tract Carcinoma
Brief Title: Pembrolizumab (MK-3475) Plus Gemcitabine/Cisplatin Versus Placebo Plus Gemcitabine/Cisplatin for First-Line Advanced and/or Unresectable Biliary Tract Carcinoma (BTC) (MK-3475-966/KEYNOTE-966)
Acronym: KEYNOTE-966
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3475-966; MK-3475-966 (Other: MSD); KEYNOTE-966 (Other: MSD); 195007 (Registry Identifier: JAPIC-CTI); 2023-506657-38 (Registry Identifier: EU CT); U1111-1294-1943 (Registry Identifier: UTN); 2019-000944-82 (EudraCT Number)
Record Dates: First submitted 2019-06-28; First posted 2019-07-01 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Biliary Tract Carcinoma
Keywords: Programmed cell death 1 (PD-1); Pembrolizumab; Cholangiocarcinoma; Gallbladder cancer; Checkpoint inhibitor; Immunotherapy; Biliary; Keytruda; Bile Duct Cancer
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body; Cholangiocarcinoma; Gallbladder Neoplasms; Bile Duct Neoplasms | interventions — pembrolizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Pembrolizumab+Gemcitabine+Cisplatin) (Experimental): Pembrolizumab, 200 mg, every 3 weeks (Q3W), Day 1 of each 3-week cycle for up to 35 cycles PLUS Gemcitabine, 1000 mg/m^2, Q3W, Day 1 and Day 8 of each cycle until progressive disease or unacceptable toxicity PLUS Cisplatin, 25 mg/m^2, Q3W, Day 1 and Day 8 of each cycle for up to 8 cycles.
  Interventions: Biological: Pembrolizumab; Drug: Gemcitabine; Drug: Cisplatin
- Arm B (Placebo+Gemcitabine+Cisplatin) (Placebo Comparator): Placebo to Pembrolizumab, 200 mg, every 3 weeks (Q3W), Day 1 of each 3-week cycle for up to 35 cycles PLUS Gemcitabine, 1000 mg/m^2, Q3W, Day 1 and Day 8 of each cycle until progressive disease or unacceptable toxicity PLUS Cisplatin, 25 mg/m^2, Q3W, Day 1 and Day 8 of each cycle for up to 8 cycles.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Placebo

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab by intravenous (IV) infusion
  Other Names: MK-3475
  Arms: Arm A (Pembrolizumab+Gemcitabine+Cisplatin)
Drug: Gemcitabine — Gemcitabine by IV infusion
  Other Names: Gemzar
Drug: Cisplatin — Cisplatin by IV infusion
  Other Names: Platinol®; Platinol®-AQ
Drug: Placebo — Placebo to pembrolizumab
  Arms: Arm B (Placebo+Gemcitabine+Cisplatin)

SUMMARY:
This is a study of pembrolizumab plus gemcitabine/cisplatin versus placebo plus gemcitabine/cisplatin as first-line therapy in participants with advanced and/or unresectable biliary tract carcinoma. The primary hypothesis is pembrolizumab plus gemcitabine/cisplatin is superior to placebo plus gemcitabine/cisplatin with respect to overall survival (OS).

ELIGIBILITY:
Inclusion Criteria

* Has histologically confirmed diagnosis of advanced (metastatic) and/or unresectable (locally advanced) biliary tract cancer (intra-or extrahepatic cholangiocarcinoma or gallbladder cancer)
* Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1), as determined by the site investigator
* Participants with a history of hepatitis B or hepatitis C can be enrolled if they meet study criteria
* Is able to provide archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion
* Has a life expectancy of greater than 3 months
* Has adequate organ function

Exclusion Criteria

* Has had previous systemic therapy for advanced (metastatic) or unresectable (locally advanced) biliary tract cancer (intra-or extra hepatic cholangiocarcinoma or gallbladder cancer)
* Has ampullary cancer
* Has small cell cancer, neuroendocrine tumors, lymphoma, sarcoma, mixed tumor histology and/or mucinous cystic neoplasms
* Has received prior therapy with an anti-programmed cell death 1 (anti-PD-1), anti- programmed cell death ligand 1 or 2 (anti-PD-L1, anti-PD-L2) agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX-40, CD137)
* Has a known history of, or any evidence of, central nervous system (CNS) metastases and/or carcinomatous meningitis, as assessed by local site investigator
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1069 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2025-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (185):
- United States (18):
  - University of Alabama at Birmingham Comprehensive Cancer Ctr ( Site 0016), Birmingham, Alabama
  - University of California San Diego Moores Cancer Center ( Site 0008), La Jolla, California
  - UCLA Hematology/Oncology - Santa Monica ( Site 0014), Los Angeles, California
  - University of California - San Francisco ( Site 0030), San Francisco, California
  - University of Colorado Hospital ( Site 0011), Aurora, Colorado
  - Hartford Hospital ( Site 0057), Hartford, Connecticut
  - Yale University ( Site 0053), New Haven, Connecticut
  - Winship Cancer Institute of Emory University ( Site 0013), Atlanta, Georgia
  - Northwest Georgia Oncology Centers PC ( Site 0045), Marietta, Georgia
  - Decatur Memorial Hospital ( Site 0056), Decatur, Illinois
  - Winthrop University Hospital ( Site 0059), Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health ( Site 0038), New York, New York
  - Columbia University/Herbert Irving Cancer Center ( Site 0009), New York, New York
  - University of Oklahoma- Stephenson Oklahoma Cancer Center ( Site 0055), Oklahoma City, Oklahoma
  - OHSU Center for Health & Healing ( Site 0044), Portland, Oregon
  - Charleston Oncology ( Site 0042), Charleston, South Carolina
  - Saint Francis Health System ( Site 0051), Greenville, South Carolina
  - Blue Ridge Cancer Care ( Site 0033), Roanoke, Virginia
- Argentina (5):
  - CEMIC ( Site 0581), Buenos Aires, Buenos Aires F.D.
  - Fundacion Favaloro ( Site 0578), Ciudad de Buenos Aires, Buenos Aires F.D.
  - Centro Medico San Roque ( Site 0579), San Miguel de Tucumán, Tucumán Province
  - Hospital Municipal de Gastroenterologia Dr. Bonorino Udaondo ( Site 0580), CABA
  - Centro Oncologico Riojano Integral ( Site 0584), La Rioja
- Australia (5):
  - Liverpool Hospital ( Site 0707), Liverpool, New South Wales
  - Mid North Coast Cancer Institute ( Site 0708), Port Macquarie, New South Wales
  - Gallipoli Medical Research Foundation ( Site 0705), Brisbane, Queensland
  - Eastern Health ( Site 0704), Box Hill, Victoria
  - Western Health-Sunshine Hospital ( Site 0709), St Albans, Victoria
- Belgium (7):
  - UZA University Hospital Antwerp ( Site 0202), Edegem, Antwerpen
  - Erasme Hospital ( Site 0204), Brussels, Bruxelles-Capitale, Region de
  - Saint-Luc UCL ( Site 0200), Brussels, Bruxelles-Capitale, Region de
  - Grand Hopital de Charleroi ( Site 0206), Charleroi, Hainaut
  - CHU de Liege ( Site 0201), Liège, Liege
  - UZ Gent ( Site 0203), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 0205), Leuven, Vlaams-Brabant
- Brazil (10):
  - Oncobio Servicos de Saude SA ( Site 0604), Nova Lima, Minas Gerais
  - Hospital de Caridade de Ijui ( Site 0602), Ijuí, Rio Grande do Sul
  - Associacao Hospitalar Moinhos de Vento ( Site 0599), Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre ( Site 0610), Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao ( Site 0601), Porto Alegre, Rio Grande do Sul
  - Instituto COI de Pesquisa Educacao e Gestao ( Site 0606), Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 0607), São Paulo
  - Hospital Paulistano - Amil Clinical Research ( Site 0603), São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia ( Site 0609), São Paulo
  - A.C. Camargo Cancer Center ( Site 0600), São Paulo
- Canada (5):
  - Tom Baker Cancer Centre ( Site 0184), Calgary, Alberta
  - Cross Cancer Institute ( Site 0183), Edmonton, Alberta
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 0182), Hamilton, Ontario
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0180), Montreal, Quebec
  - McGill University Health Centre ( Site 0179), Montreal, Quebec
- Chile (6):
  - IC La Serena Research ( Site 0630), La Serena, Coquimbo Region
  - Servicios Medicos Urumed ( Site 0621), Rancagua, Lbtdr Gen Bernardo O Higgins
  - Fundacion Arturo Lopez Perez FALP ( Site 0623), Santiago, Region M. de Santiago
  - Sociedad Oncovida S.A. ( Site 0626), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0620), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 0622), Temuco, Región de la Araucanía
- China (22):
  - Anhui Provincial Hospital ( Site 0140), Hefei, Anhui
  - Beijing Cancer Hospital ( Site 0138), Beijing, Beijing Municipality
  - Peking Union Medical College Hospital ( Site 0150), Beijing, Beijing Municipality
  - First Affiliated Hospital of The Third Military Medical University ( Site 0130), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 0154), Fuzhou, Fujian
  - 900 Hospital of the Joint ( Site 0137), Fuzhou, Fujian
  - Guangdong Provincial People s Hospital ( Site 0161), Guangzhou, Guangdong
  - The Third Xiangya Hospital of Central South University ( Site 0157), Changsha, Hainan
  - Harbin Medical University Cancer Hospital ( Site 0133), Harbin, Heilongjiang
  - Hunan Provincial People Hospital ( Site 0142), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 0132), Changsha, Hunan
  - The 81st Hospital of PLA ( Site 0128), Nanjing, Jiangsu
  - The First Hospital of Jilin University ( Site 0131), Changchun, Jilin
  - Zhongshan Hospital Fudan University ( Site 0129), Shanghai, Shanghai Municipality
  - Renji Hospital Shanghai Jiaotong University School of Medicine ( Site 0158), Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center ( Site 0160), Shanghai, Shanghai Municipality
  - Tangdu Hospital ( Site 0146), Xi’an, Shanxi
  - The First Affiliated Hospital of Xi an Jiaotong University ( Site 0145), Xi’an, Shanxi
  - West China Hospital of Sichuan University ( Site 0147), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital ( Site 0155), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital Zhejiang University ( Site 0136), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0134), Hangzhou, Zhejiang
- France (6):
  - CHU Bordeaux Haut-Leveque Centre Francois Magendie ( Site 0245), Pessac, Gironde
  - A.P.H. Paris, Hopital Beaujon ( Site 0247), Clichy, Hauts-de-Seine
  - CHU de Montpellier - Hopital Saint-Eloi ( Site 0248), Montpellier, Herault
  - Centre Eugene Marquis ( Site 0242), Rennes, Ille-et-Vilaine
  - CHU Clermont-Ferrand - Site Estaing ( Site 0249), Clermont-Ferrand, Puy-de-Dome
  - Gustave Roussy ( Site 0244), Villejuif, Val-de-Marne
- Germany (11):
  - Universitaetsklinikum Ulm ( Site 0267), Ulm, Baden-Wurttemberg
  - Klinikum der Ludwig - Maximilian Universitat Munchen ( Site 0264), Munich, Bavaria
  - Krankenhaus Nordwest ( Site 0266), Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover ( Site 0265), Hanover, Lower Saxony
  - Universitaetsklinikum Aachen AOER ( Site 0275), Aachen, North Rhine-Westphalia
  - Universitaetsklinikum Koeln ( Site 0274), Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Essen ( Site 0273), Essen, North Rhine-Westphalia
  - Staedtisches Klinikum Dresden ( Site 0272), Dresden, Saxony
  - Universitaetsklinikum Magdeburg A.o.R. ( Site 0271), Magdeburg, Saxony-Anhalt
  - Charite - Universtitatsmedizin Berlin CCM ( Site 0269), Berlin
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 0268), Hamburg
- Hong Kong (5):
  - Pamela Youde Nethersole Eastern Hospital ( Site 0857), Hong Kong
  - Prince of Wales Hospital ( Site 0855), Hong Kong
  - Princess Margaret Hospital. ( Site 0856), Hong Kong
  - Queen Mary Hospital ( Site 0851), Hong Kong
  - Queen Elizabeth Hospital. ( Site 0854), Kowloon
- Ireland (4):
  - Cork University Hospital ( Site 0538), Cork
  - Bon Secours Hospital ( Site 0526), Cork
  - Tallaght University Hospital ( Site 0522), Dublin
  - St Vincents University Hospital ( Site 0521), Dublin
- Israel (4):
  - Rambam Medical Center ( Site 0308), Haifa
  - Hadassah Ein Karem - Sharett Institute of Oncology ( Site 0309), Jerusalem
  - Rabin Medical Center ( Site 0307), Petah Tikva
  - Sourasky Medical Center ( Site 0306), Tel Aviv
- Italy (7):
  - Universita Cattolica del Sacro Cuore - Policlinico Gemelli ( Site 0329), Rome, Abruzzo
  - Policlinico S. Orsola-Malpighi ( Site 0333), Bologna
  - A.O. di Rilievo Nazionale e di alta Specializzazione Garibaldi ( Site 0330), Catania
  - ASST Grande Ospedale Metropolitano Niguarda ( Site 0332), Milan
  - Azienda Ospedaliero Universitaria Pisana ( Site 0326), Pisa
  - Policlinico Universitario Campus Biomedico ( Site 0328), Roma
  - Azienda Ospedaliera Universitaria di Verona ( Site 0334), Verona
- Japan (11):
  - Aichi Cancer Center Hospital ( Site 0080), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 0081), Kashiwa, Chiba
  - Kobe City Medical Center General Hospital ( Site 0087), Kobe, Hyōgo
  - Kagawa University Hospital ( Site 0086), Kita-gun, Kagawa-ken
  - Kanagawa Cancer Center ( Site 0079), Yokohama, Kanagawa
  - Osaka University Hospital ( Site 0085), Suita, Osaka
  - Kyorin University Hospital ( Site 0077), Mitaka, Tokyo
  - National Hospital Organization Kyushu Cancer Center ( Site 0078), Fukuoka
  - Kyoto University Hospital ( Site 0083), Kyoto
  - Osaka International Cancer Institute ( Site 0084), Osaka
  - The Cancer Institute Hospital of JFCR ( Site 0082), Tokyo
- Malaysia (6):
  - Hospital Sultan Ismail ( Site 0772), Johor Bahru, Johor
  - University Malaya Medical Centre ( Site 0770), Lembah Pantai, Kuala Lumpur
  - Hospital Pulau Pinang ( Site 0773), George Town, Pulau Pinang
  - Institut Kanser Negara - National Cancer Institute ( Site 0767), Putrajaya, Putrajaya
  - Hospital Kuala Lumpur ( Site 0768), Kuala Lumpur
  - Pantai Hospital Kuala Lumpur ( Site 0771), Kuala Lumpur
- Netherlands (5):
  - Maastricht University Medical Centre ( Site 0347), Maastricht, Limburg
  - AMC ( Site 0348), Amsterdam, North Holland
  - Erasmus University Medical Center ( Site 0352), Rotterdam, South Holland
  - UMCG ( Site 0349), Groningen
  - Universitair Medisch Centrum Utrecht ( Site 0351), Utrecht
- Auckland City Hospital ( Site 0725), Auckland, New Zealand
- South Korea (11):
  - Chonnam National University Hwasun Hospital ( Site 0837), Hwasun Gun, Jeonranamdo
  - CHA Bundang Medical Center CHA University ( Site 0835), Seongnam, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 0833), Seongnam-si, Kyonggi-do
  - Ajou University Hospital, Clinical Research Center ( Site 0838), Suwon, Kyonggi-do
  - Kyungpook National University Chilgok Hospital ( Site 0834), Daegu, Taegu-Kwangyokshi
  - Chungnam National University Hospital ( Site 0840), Daejeon, Taejon-Kwangyokshi
  - Severance Hospital Yonsei University Health System ( Site 0836), Seoul
  - Asan Medical Center ( Site 0830), Seoul
  - Samsung Medical Center ( Site 0831), Seoul
  - The Catholic University of Korea. Seoul St. Mary s Hospital ( Site 0839), Seoul
  - Korea University Guro Hospital ( Site 0832), Seoul
- Spain (5):
  - Hospital Universitario General de Asturias ( Site 0434), Oviedo, Principality of Asturias
  - Hospital General Universitari Vall d Hebron ( Site 0432), Barcelona
  - Hospital General Universitario Gregorio Maranon ( Site 0433), Madrid
  - Hospital Universitario HM Sanchinarro ( Site 0435), Madrid
  - Hospital Regional Universitario Carlos Haya ( Site 0431), Málaga
- Taiwan (7):
  - Taipei Veterans General Hospital ( Site 0861), Taipei,, Taipei
  - Chang Gung Medical Foundation. Kaohsiung Branch ( Site 0865), Kaohsiung City
  - China Medical University Hospital ( Site 0862), Taichung
  - National Cheng Kung University Hospital ( Site 0864), Tainan
  - National Taiwan University Hospital ( Site 0860), Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center ( Site 0863), Taipei
  - Chang Gung Medical Foundation. Linkou ( Site 0853), Taoyuan District
- Thailand (7):
  - King Chulalongkorn Memorial Hospital ( Site 0884), Bangkok, Bangkok
  - Ramathibodi Hospital. ( Site 0889), Bangkok, Bangkok
  - Siriraj Hospital ( Site 0888), Bangkok, Bangkok
  - Sunpasithiprasong Hospital ( Site 0883), Ubonratchathani, Changwat Ubon Ratchathani
  - Maharaj Nakorn Chiang Mai Hospital ( Site 0887), Chiang Mai
  - Srinagarind Hospital ( Site 0885), Khon Kaen
  - Udon Thani Cancer Hospital ( Site 0886), Udon Thani
- Turkey (Türkiye) (9):
  - Inonu Universitesi Medical Fakultesi ( Site 0501), Malatya, Adana
  - Baskent University Adana Training Hospital ( Site 0499), Adana
  - Hacettepe University Faculty of Medicine ( Site 0498), Ankara
  - Abdurrahman Yurtaslan Onkoloji Hastanesi ( Site 0494), Ankara
  - Gazi Universitesi Tip Fakultesi ( Site 0496), Ankara
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 0506), Istanbul
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi-oncology ( Site 0495), Istanbul
  - Izmir Medical Park Hospital Department of Medical Oncology ( Site 0502), Izmir
  - Erciyes Universitesi Tip Fakultesi ( Site 0500), Kayseri
- United Kingdom (8):
  - Aberdeen Royal Infirmary ( Site 0529), Aberdeen, Aberdeen City
  - Royal Free London NHS Foundation Trust ( Site 0520), London, London, City of
  - Royal Marsden Hospital ( Site 0536), London, London, City of
  - Imperial College Healthcare NHS Trust - Hammersmith Hospital ( Site 0525), London, London, City of
  - Royal Marsden NHS Foundation Trust ( Site 0535), Sutton, Surrey
  - Belfast City Hospital ( Site 0517), Belfast
  - University Hospital Coventry and Warwickshire NHS Trust ( Site 0518), Coventry
  - The Christie NHS Foundation Trust ( Site 0537), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Kelley RK, Ueno M, Yoo C, Finn RS, Furuse J, Ren Z, Yau T, Klumpen HJ, Chan SL, Ozaka M, Verslype C, Bouattour M, Park JO, Barajas O, Pelzer U, Valle JW, Yu L, Malhotra U, Siegel AB, Edeline J, Vogel A; KEYNOTE-966 Investigators. Pembrolizumab in combination with gemcitabine and cisplatin compared with gemcitabine and cisplatin alone for patients with advanced biliary tract cancer (KEYNOTE-966): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2023 Jun 3;401(10391):1853-1865. doi: 10.1016/S0140-6736(23)00727-4. Epub 2023 Apr 16. PMID 37075781
- [Derived] Jiang C, Zhou K, Shu P. Cost-effectiveness analysis of pembrolizumab plus chemotherapy as first-line treatment for advanced biliary tract cancer: perspectives from US and Chinese payers. BMJ Open. 2025 Apr 23;15(4):e094047. doi: 10.1136/bmjopen-2024-094047. PMID 40268484
- [Derived] Luo X, Cai T, Wu J, Li X, Wang X, Ma H. Cost-effectiveness of pembrolizumab plus chemotherapy vs. chemotherapy as first-line treatment for advanced biliary tract cancer in China and the US. Front Pharmacol. 2024 Aug 14;15:1393559. doi: 10.3389/fphar.2024.1393559. eCollection 2024. PMID 39206260
- [Derived] Keller HR, Fluke L, Forrester JA, Wolf RF. Identifying Indications for Neoadjuvant Therapy in Cholangiocarcinoma. Oncology (Williston Park). 2024 Apr 11;38(4):160-162. doi: 10.46883/2024.25921017. PMID 38661512
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26256&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As of the data cut-off (DCO) (15-DEC-2022) for the final analysis (FA), a total of 1069 participants were randomized to the Intent-to-Treat (ITT) population (533 in the pembrolizumab plus chemotherapy group and 536 in the placebo plus chemotherapy group)
Groups:
- Arm A (Pembrolizumab+Gemcitabine+Cisplatin): Pembrolizumab, 200 mg, every 3 weeks (Q3W), Day 1 of each 3-week cycle for up to 35 cycles PLUS Gemcitabine, 1000 mg/m^2, Q3W, Day 1 and Day 8 of each cycle until progressive disease or unacceptable toxicity plus Cisplatin, 25 mg/m^2, Q3W, Day 1 and Day 8 of each cycle for up to 8 cycles. Participants in Arm A who stopped study intervention after achieving stable-disease (SD) or better may have been eligible to receive additional pembrolizumab for up to 17 cycles if they experienced radiographic disease progression while off study intervention, according to the protocol-defined criteria. Gemcitabine may have been continued until progressive disease (PD) or unacceptable toxicity during second course at investigator's discretion.
Period: Overall Study
Arm/Group | Arm A (Pembrolizumab+Gemcitabine+Cisplatin) | Arm B (Placebo+Gemcitabine+Cisplatin)
Started | 533 | 536
Completed | 0 | 0
Not Completed | 533 | 536
Not completed — Death | 409 | 443
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Participant On-going | 119 | 90

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Pembrolizumab+Gemcitabine+Cisplatin) | Arm B (Placebo+Gemcitabine+Cisplatin) | Total
Number analyzed (Participants) | 533 | 536 | 1069
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (10.3) | 61.8 (11.0) | 62.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 253 | 264 | 517
  Male | 280 | 272 | 552
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 52 | 111
  Not Hispanic or Latino | 433 | 449 | 882
  Unknown or Not Reported | 41 | 35 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 245 | 250 | 495
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 11 | 3 | 14
  White | 256 | 268 | 524
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 13 | 12 | 25
Geographic Region [Number; unit: Number of Participants]
  Asian | 242 | 244 | 486
  Non-Asian | 291 | 292 | 583
Disease Status [Number; unit: Participants]
  Locally Advanced | 60 | 66 | 126
  Metastatic | 473 | 470 | 943
Site of Origin [Number; unit: Participants]
  Gallbladder | 115 | 118 | 233
  Intrahepatic | 320 | 313 | 633
  Extrahepatic | 98 | 105 | 203

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from randomization to death due to any cause.
Time Frame: Up to approximately 38 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Pembrolizumab+Gemcitabine+Cisplatin) | Arm B (Placebo+Gemcitabine+Cisplatin)
Number analyzed (Participants) | 533 | 536
Months | 12.7 [11.5 to 13.6] | 10.9 [9.9 to 11.6]
Statistical Analysis 1: Comparison: Arm A (Pembrolizumab+Gemcitabine+Cisplatin) vs Arm B (Placebo+Gemcitabine+Cisplatin); Test type: Superiority; p = 0.0034, Regression, Cox; One-sided p-value based on log-rank test stratified by geographic region, disease status, site of origin with small strata collapsed; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.72 to 0.95] — HR=Arm A/Arm B

2. Secondary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (BICR)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 by BICR, or death due to any cause, whichever occurred first.
Time Frame: Up to approximately 26 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Pembrolizumab+Gemcitabine+Cisplatin) | Arm B (Placebo+Gemcitabine+Cisplatin)
Number analyzed (Participants) | 533 | 536
Months | 6.5 [5.7 to 6.9] | 5.6 [5.1 to 6.6]
Statistical Analysis 1: Comparison: Arm A (Pembrolizumab+Gemcitabine+Cisplatin) vs Arm B (Placebo+Gemcitabine+Cisplatin); Test type: Superiority; p = 0.0225, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.75 to 1.00] — HR=Arm A/Arm B

3. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: ORR was defined as the percentage of participants who have a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: a ≥30% decrease in the sum of diameters [SOD] of target lesions) as assessed by BICR per RECIST 1.1, which was adjusted for this study to allow a maximum of 10 target lesions in total and 5 per organ.
Time Frame: Up to approximately 26 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A (Pembrolizumab+Gemcitabine+Cisplatin) | Arm B (Placebo+Gemcitabine+Cisplatin)
Number analyzed (Participants) | 533 | 536
Percentage of Participants | 28.7 [24.9 to 32.8] | 28.5 [24.8 to 32.6]
Statistical Analysis 1: Comparison: Arm A (Pembrolizumab+Gemcitabine+Cisplatin) vs Arm B (Placebo+Gemcitabine+Cisplatin); Test type: Superiority; p = 0.4735, Miettinen & Nurminen — One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentages = 0.2, 95% CI 2-sided [-5.2 to 5.6] — Difference=Arm A minus Arm B

4. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR
Description: For participants who demonstrate a confirmed CR or PR, DOR was the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurred first.
Time Frame: Up to approximately 38 months
Population: All randomized participants with CR or PR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Pembrolizumab+Gemcitabine+Cisplatin) | Arm B (Placebo+Gemcitabine+Cisplatin)
Number analyzed (Participants) | 153 | 153
Months | 9.7 [1.2 to 22.7] | 6.9 [0.0 to 19.2]

5. Secondary Outcome: Number of Participants Who Experience One or More Adverse Events (AE)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it was considered related to the medical treatment or procedure, that occurred during the course of the study.
Time Frame: Up to approximately 38 months
Population: All Participants as Treated (APaT) population, which consisted of all randomized participants who received at least 1 dose of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Pembrolizumab+Gemcitabine+Cisplatin) | Arm B (Placebo+Gemcitabine+Cisplatin)
Number analyzed (Participants) | 529 | 534
Participants | 524 | 532

6. Secondary Outcome: Number of Participants Who Discontinued Study Intervention Due to an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it was considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to approximately 38 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Pembrolizumab+Gemcitabine+Cisplatin) | Arm B (Placebo+Gemcitabine+Cisplatin)
Number analyzed (Participants) | 529 | 534
Participants | 138 | 122

ADVERSE EVENTS:
Time Frame: Up to approximately 38 months
Description: All-Cause Mortality included all allocated participants. Serious and Other AEs were reported according to treatment course for all participants who received ≥1 dose of study treatment.
Groups:
- Pembrolizumab + Chemotherapy: Pembrolizumab, 200 mg, every 3 weeks (Q3W), Day 1 of each 3-week cycle for up to 35 cycles PLUS Gemcitabine, 1000 mg/m^2, Q3W, Day 1 and Day 8 of each cycle until progressive disease or unacceptable toxicity plus Cisplatin, 25 mg/m^2, Q3W, Day 1 and Day 8 of each cycle for up to 8 cycles.
- Placebo + Chemotherapy: Placebo to Pembrolizumab, 200 mg, every 3 weeks (Q3W), Day 1 of each 3-week cycle for up to 35 cycles PLUS Gemcitabine, 1000 mg/m^2, Q3W, Day 1 and Day 8 of each cycle until progressive disease or unacceptable toxicity PLUS Cisplatin, 25 mg/m^2, Q3W, Day 1 and Day 8 of each cycle for up to 8 cycles.
- Pembrolizumab Second Course: Participants in Arm A who stopped study intervention after achieving stable-disease (SD) or better may have been eligible to receive additional pembrolizumab for up to 17 cycles if they experienced radiographic disease progression while off study intervention, according to the protocol-defined criteria. Gemcitabine may have been continued until progressive disease (PD) or unacceptable toxicity during second course at investigator's discretion.
Arm/Group | Pembrolizumab + Chemotherapy | Placebo + Chemotherapy | Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 413/533 | 443/536 | 1/2
Serious Adverse Events (participants affected / at risk) | 276/529 | 263/534 | 0/2
Other Adverse Events (participants affected / at risk) | 512/529 | 522/534 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Chemotherapy (N=529) | Placebo + Chemotherapy (N=534) | Pembrolizumab Second Course (N=2)
Anaemia (Blood and lymphatic system disorders) | 13 (13) | 10 (10) | 0 (0)
Coombs negative haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (8) | 8 (8) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 6 (6) | 3 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 7 (7) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 6 (7) | 13 (14) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 6 (6) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Fistula of small intestine (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 4 (4) | 4 (6) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Intestinal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pancreatolithiasis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Prepyloric stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (7) | 4 (4) | 0 (0)
Asthenia (General disorders) | 2 (3) | 3 (3) | 0 (0)
Death (General disorders) | 3 (3) | 5 (5) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperpyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Puncture site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 30 (34) | 12 (15) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 12 (14) | 16 (18) | 0 (0)
Biloma (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 31 (39) | 24 (38) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 7 (8) | 3 (3) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 3 (3) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatic displacement (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic ischaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 3 (3) | 4 (4) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 3 (3) | 5 (6) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion related hypersensitivity reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 8 (8) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Biliary tract infection (Infections and infestations) | 17 (21) | 18 (25) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Burkholderia cepacia complex infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 7 (7) | 8 (8) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 6 (6) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cholangitis infective (Infections and infestations) | 0 (0) | 3 (4) | 0 (0)
Device related infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fungal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 4 (4) | 11 (13) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 4 (4) | 3 (3) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 8 (9) | 8 (9) | 0 (0)
Pneumonia acinetobacter (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 13 (15) | 16 (17) | 0 (0)
Septic embolus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Spontaneous bacterial peritonitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 10 (10) | 6 (6) | 0 (0)
Urosepsis (Infections and infestations) | 1 (2) | 2 (2) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative adhesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stoma site ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ureteric injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 4 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 5 (5) | 4 (4) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 11 (13) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 19 (19) | 10 (12) | 0 (0)
Transaminases increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Food refusal (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Benign neoplasm of testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 5 (5) | 4 (4) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Radicular pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 2 (3) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 2 (2) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (5) | 10 (12) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (3) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Renal vein thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 8 (8) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Euthanasia (Surgical and medical procedures) | 2 (2) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Inferior vena caval occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Vena cava embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Chemotherapy (N=529) | Placebo + Chemotherapy (N=534) | Pembrolizumab Second Course (N=2)
Anaemia (Blood and lymphatic system disorders) | 315 (528) | 306 (486) | 0 (0)
Hypothyroidism (Endocrine disorders) | 45 (46) | 14 (14) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 37 (41) | 34 (43) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 88 (122) | 117 (152) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 40 (53) | 56 (72) | 0 (0)
Ascites (Gastrointestinal disorders) | 29 (31) | 33 (34) | 0 (0)
Constipation (Gastrointestinal disorders) | 185 (227) | 188 (233) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 102 (149) | 93 (149) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 33 (36) | 55 (64) | 1 (1)
Nausea (Gastrointestinal disorders) | 232 (418) | 245 (421) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 26 (30) | 34 (37) | 1 (1)
Vomiting (Gastrointestinal disorders) | 120 (234) | 127 (268) | 0 (0)
Asthenia (General disorders) | 75 (134) | 93 (165) | 0 (0)
Fatigue (General disorders) | 186 (281) | 170 (231) | 0 (0)
Malaise (General disorders) | 36 (65) | 31 (59) | 0 (0)
Mucosal inflammation (General disorders) | 28 (34) | 23 (31) | 0 (0)
Oedema peripheral (General disorders) | 73 (87) | 85 (124) | 0 (0)
Pyrexia (General disorders) | 118 (228) | 96 (172) | 0 (0)
Urinary tract infection (Infections and infestations) | 29 (37) | 23 (26) | 0 (0)
Alanine aminotransferase increased (Investigations) | 86 (142) | 110 (169) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 88 (160) | 98 (187) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 42 (59) | 52 (72) | 0 (0)
Blood bilirubin increased (Investigations) | 46 (69) | 61 (80) | 0 (0)
Blood creatinine increased (Investigations) | 56 (101) | 58 (103) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 23 (30) | 29 (39) | 0 (0)
Lymphocyte count decreased (Investigations) | 23 (49) | 29 (48) | 0 (0)
Neutrophil count decreased (Investigations) | 328 (1386) | 327 (1269) | 0 (0)
Platelet count decreased (Investigations) | 207 (571) | 211 (568) | 0 (0)
Weight decreased (Investigations) | 51 (52) | 63 (75) | 0 (0)
White blood cell count decreased (Investigations) | 141 (740) | 127 (616) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 141 (185) | 151 (206) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 36 (58) | 40 (51) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 35 (78) | 29 (35) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 38 (52) | 49 (67) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 48 (67) | 67 (92) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 79 (148) | 79 (139) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 51 (86) | 49 (59) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 (45) | 41 (50) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 53 (65) | 72 (77) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 27 (36) | 30 (33) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 (35) | 22 (24) | 0 (0)
Dizziness (Nervous system disorders) | 32 (44) | 50 (55) | 1 (1)
Dysgeusia (Nervous system disorders) | 31 (34) | 32 (34) | 0 (0)
Headache (Nervous system disorders) | 53 (79) | 45 (53) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 21 (23) | 29 (31) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 31 (33) | 29 (30) | 0 (0)
Insomnia (Psychiatric disorders) | 41 (46) | 41 (45) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 36 (42) | 37 (43) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 51 (59) | 51 (56) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 55 (58) | 68 (71) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 77 (106) | 51 (60) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 88 (113) | 49 (64) | 0 (0)
Hypertension (Vascular disorders) | 34 (40) | 37 (60) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT04003636/Prot_SAP_000.pdf